CLINICAL TRIAL: NCT01096108
Title: Enhancing Quit and Win Contests to Improve Smoking Cessation Among College Students
Brief Title: Quit and Win Contests to Improve Smoking Cessation Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 2008NTLS155; 0901S57761 (Other: IRB, University of Minnesota); R01 HL093114-01 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Tobacco Use Cessation
Keywords: Smoking cessation; Quit smoking; Quit & Win
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Contest (Experimental): Smoking abstinence, 1 prize award (month 1)
  Interventions: Behavioral: Standard contest (1 month)
- Standard Contest plus MAPS (Experimental): Smoking abstinence, 1 prize award (month 1) plus motivational and problem-solving counseling (MAPS - Counseling phone calls); 20 weeks.
  Interventions: Behavioral: Standard contest (1 month); Behavioral: Motivational and Problem-Solving
- Extended Contests (Experimental): Smoking abstinence, 3 contest prize awards (contests 1, 2 and 3)
  Interventions: Behavioral: Extended Contests
- Extended Contests plus MAPS (Experimental): Extended quit and win contests (3 successive monthly contests) plus motivational and problem-solving counseling (MAPS). {Smoking abstinence, 3 contest prize awards (contests 1, 2 and 3) plus Counseling phone calls.
  Interventions: Behavioral: Motivational and Problem-Solving; Behavioral: Extended Contests

INTERVENTIONS:
Behavioral: Standard contest (1 month) — Smoking abstinence, 1 prize award (month 1)
  Arms: Standard Contest; Standard Contest plus MAPS
Behavioral: Motivational and Problem-Solving — Counseling phone calls
  Arms: Extended Contests plus MAPS; Standard Contest plus MAPS
Behavioral: Extended Contests — Smoking abstinence, 3 contest prize awards (contests 1, 2 and 3)
  Arms: Extended Contests; Extended Contests plus MAPS

SUMMARY:
Standard Quit and Win contests, in which smokers typically quit for one month in return for the opportunity to win prizes, are simple and easy to implement and may be cost-effective in encouraging smokers to quit. By extending contest length and enhancing counseling content, Quit and Win contests may be more effective at encouraging smoking abstinence.

This study aims to evaluate the efficacy of extended and content-enhanced Quit and Win contests to enhance smoking abstinence at college campuses.

DETAILED DESCRIPTION:
Participants will be randomized to 1 of 4 treatment groups with varying counseling treatments and contest lengths. All participants receive a 2 week supply of nicotine replacement therapy (NRT) and weekly support emails. Follow-up assessment surveys occur at 1, 3, 4 and 6 months post enrollment.

Participants who have completed the follow-up assessment surveys and self-reported that they are tobacco-free will be asked to provide a urine sample in order to verify abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled full or part-time at one of the participating campuses
* Smoke at least 10 days per month
* Intending to be in school for the entire academic year (i.e., next 2 semesters)
* Willing to provide a baseline urine sample to verify smoking status
* Able to read English
* Access to working telephone for phone-based counseling and surveys
* Access to a computer with internet access
* Provide written informed consent

Exclusion Criteria:

* Prior to concurrent enrollment in this study through a different college campus or in a different academic year
* those who have used a cessation aid within the last 7 days
* pregnant or planning to become pregnant in next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1318 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of extended versus standard quit and win contests | 6 Months
  The aim is to evaluate the separate and combined efficacy of increased dose of treatment and adding counseling to enhance smoking abstinence among college students

SECONDARY OUTCOMES:
Efficacy of motivational and problem solving counseling versus no counseling | 6 Months
  The aim is to 1) determine relative cost-effectiveness of extended incentives and motivational and problem-solving (MAPS) counseling. 2) Examine potential mediators and moderators of intervention effects.

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Thomas, Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Thomas JL, Bengtson JE, Wang Q, Luo X, Marigi E, Ghidei W, Ahluwalia JS. Abstinence rates among college cigarette smokers enrolled in a randomized clinical trial evaluating Quit and Win contests: The impact of concurrent hookah use. Prev Med. 2015 Jul;76:20-5. doi: 10.1016/j.ypmed.2015.03.010. Epub 2015 Mar 13. PMID 25773472